CLINICAL TRIAL: NCT04087161
Title: Multicenter Assessment of a Bedside-testing System (Nephrocheck™) for Acute Kidney Injury After Thoracoabdominal Aortic Surgery
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Collaborators: Münster, University Hospital, Department of Vascular Surgery (Unknown); Berlin, University medicine Charité, Department of Vascular Surgery (Unknown)
Responsible Party: Principal Investigator, Alexander Gombert, Prinicipal Investigator, RWTH Aachen University
Other Study IDs: 29012015
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Early Assessment of AKI After TAAA Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Other: Nephrocheck bed side testing of AKI — Usage of Nephrocheck system to assess AKI after open TAAA repair

SUMMARY:
Assessment of postoperative acute kidney insufficiency according to the KDIGO classification using the Nephrocheck system.

Multicentric, prospective study Open TAAA Repair in 3-4 centers in Germany and Europe

ELIGIBILITY:
Inclusion Criteria:

elective open TAAA repai

18-80 years

no pregnancy

Exclusion Criteria:

emergency treatment participation in another Trial renal replacement therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective, open TAAA repair
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury after open TAAA repair | 90 days after surgery
  Acute kidney injury defined according to the KDIGO classification and its association with the Nephrocheck assessment results

SECONDARY OUTCOMES:
Mortality, major adverse events such as any complication | 90 days after surgery
  Any severe adverse Outcome after open TAAA repair and its association with the Nephrocheck assessment results

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Doukas P, Frese JP, Eierhoff T, Hellfritsch G, Raude B, Jacobs MJ, Greiner A, Oberhuber A, Gombert A. The NephroCheck bedside system for detecting stage 3 acute kidney injury after open thoracoabdominal aortic repair. Sci Rep. 2023 Jul 9;13(1):11096. doi: 10.1038/s41598-023-38242-2. PMID 37423933